CLINICAL TRIAL: NCT05121155
Title: Brain Skull Deformation as a Non-invasive Intracranial Pressure (ICP) Measure: Comparison Between Invasive and Noninvasive Methods.
Brief Title: Brain Skull Deformation as a Non-invasive Intracranial Pressure (ICP) Measure
Status: Completed | Type: Observational
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Gisele Sampaio Silva, Profa. Dra Gisele Sampaio Silva, Federal University of São Paulo
Other Study IDs: 03843118.0.0000.5505
Record Dates: First submitted 2021-10-24; First posted 2021-11-16 (Actual); Last update posted 2021-11-16 (Actual); Status verified 2021-11

CONDITIONS: Subarachnoid Hemorrhage; Stroke; Stroke, Ischemic; Stroke Hemorrhagic; Intracranial Hypertension
Keywords: non invasive icp monitor; icp wave morphology
MeSH Terms: conditions — Subarachnoid Hemorrhage; Stroke; Ischemic Stroke; Hemorrhagic Stroke; Intracranial Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

INTERVENTIONS:
Device: ICP wave morphology comparison between a non-invasive (Brain4care) and a invasive method — We prospectively collected data of adults admitted to an intensive care unit (ICU) with subarachnoid hemorrhage (SAH), intracerebral hemorrhage (ICH) or ischemic stroke (IS) in whom invasive ICP monitoring placed. Measures had been simultaneously collected from the following non-invasive indices: optic nerve sheath diameter (ONSD), pulsatility index (PI) using transcranial Doppler (TCD), a 5-point visual scale designed for Computed Tomography (CT) and two parameters (time-to-peak [TTP] and P2/P1 ratio) of a non-invasive ICP wave morphology monitor (Brain4care[B4c]). Intracranial hypertension was defined as an invasively measured ICP > 20 mmHg for at least five minutes
  Other Names: Estimation of Intracranial Hypertension using non-invasive methods

SUMMARY:
Background: Although placement of an intra-cerebral catheter remains the gold standard method for measuring intracranial pressure (ICP), there are several limitations to the method. Objectives: The main objective of this study was to compare the correlation and the agreement of the wave morphology between the ICP (standard ICP monitoring) and a new nICP monitor in patients admitted with stroke. Our secondary objective was to estimate the accuracy of four non-invasive methods to assess intracranial hypertension. Methods: We prospectively collected data of adults admitted to an intensive care unit (ICU) with subarachnoid hemorrhage (SAH), intracerebral hemorrhage (ICH) or ischemic stroke (IS) in whom invasive ICP monitoring placed. Measures had been simultaneously collected from the following non-invasive indices: optic nerve sheath diameter (ONSD), pulsatility index (PI) using transcranial Doppler (TCD), a 5-point visual scale designed for Computed Tomography (CT) and two parameters (time-to-peak [TTP] and P2/P1 ratio) of a non-invasive ICP wave morphology monitor (Brain4care[B4c]). Intracranial hypertension was defined as an invasively measured ICP > 20 mmHg for at least five minutes.

ELIGIBILITY:
Inclusion Criteria:

- Adult inpatients from a dedicated neurological intensive care unit with ischemic (IS) or hemorrhagic stroke who needed invasive ICP monitoring were prospectively evaluated from March 2019 to March 2020 (before the COVID-19 pandemic).

Exclusion Criteria:

* We excluded patients with chronic neurological diseases (demyelinating diseases, chronic hydrocephalus, pseudotumor brain), suspected brain death, and patients monitored with non-ventricular sensors (e.g., subdural or epidural).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: From a total of 30 patients with invasive ICP monitor evaluated in our hospital between March 2019 and March 2020 (pre-Covid-19), 18 patients fulfilled inclusion and exclusion criteria. A total of 60 monitorizations were performed. We included 14 patients with subarachnoid hemorrhage (SAH), one with IS, and three with ICH. All SAH were aneurysmatic, all ICH were hypertensives and the only IS was a cardioembolic malignant middle cerebral artery stroke. There were no side effects from the use of the noninvasive method.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Comparison between ICP morphology between a non invasive (Brain4care [B4c]) and a invasive (intraventricular) method | At least 30 minutes for every patient
  Parameter of the ICP wave between methods were compared (P2/P1 ratio)
Comparison between ICP morphology between a non invasive (Brain4care [B4c]) and a invasive (intraventricular) method | At least 30 minutes for every patient
  Parameter of the ICP wave between methods were compared (Time-to-Peak)

SECONDARY OUTCOMES:
Estimation of Intracranial Hypertension using Transcranial Doppler | At least 5 minutes after EVD closure
  We measured the Pulsatility Index using transcranial Doppler (TCD) and calculated a ROC curve to calculate its discriminatory power
Estimation of Intracranial Hypertension using optic nerve sheath diameter (ONSD) | At least 5 minutes after EVD closure
  We measured the ONSD for both eyes and calculated a ROC curve to evaluate its discriminatory power in detecting Intracranial Hypertension
Estimation of Intracranial Hypertension using a non-invasive ICP wave parameter (P2/P1 ratio). | At least 5 minutes after EVD closure
  We measured the mean P2/P1 ratio and calculated a ROC curve to evaluate its discriminatory power in detecting Intracranial Hypertension.
  We calculated the points in the scale and built a ROC curve to evaluate its discriminatory power in detecting Intracranial Hypertension
Estimation of Intracranial Hypertension using a non-invasive ICP wave parameter (Time-to_peak). | At least 5 minutes after EVD closure
  We measured the mean TTP and calculated a ROC curve to evaluate its discriminatory power in detecting Intracranial Hypertension.
Estimation of Intracranial Hypertension using a 5-point visual scale designed for Computed Tomography (CT) | At least 5 minutes after EVD closure
  We calculated the points in the scale and built a ROC curve to evaluate its discriminatory power in detecting Intracranial Hypertension

CONTACTS AND LOCATIONS:
Locations (1):
- Federal University of São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
As soon as the data are published, we intend to share it.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Result] Moraes FM, Silva GS. Noninvasive intracranial pressure monitoring methods: a critical review. Arq Neuropsiquiatr. 2021 May;79(5):437-446. doi: 10.1590/0004-282X-ANP-2020-0300. PMID 34161530
- [Derived] de Moraes FM, Brasil S, Frigieri G, Robba C, Paiva W, Silva GS. ICP wave morphology as a screening test to exclude intracranial hypertension in brain-injured patients: a non-invasive perspective. J Clin Monit Comput. 2024 Aug;38(4):773-782. doi: 10.1007/s10877-023-01120-3. Epub 2024 Feb 14. PMID 38355918
- [Derived] de Moraes FM, Rocha E, Barros FCD, Freitas FGR, Miranda M, Valiente RA, de Andrade JBC, Neto FEAC, Silva GS. Waveform Morphology as a Surrogate for ICP Monitoring: A Comparison Between an Invasive and a Noninvasive Method. Neurocrit Care. 2022 Aug;37(1):219-227. doi: 10.1007/s12028-022-01477-4. Epub 2022 Mar 24. PMID 35332426